CLINICAL TRIAL: NCT05156112
Title: Examining Early Intervention Obstructive Sleep Apnea Treatment on Long-Term Outcomes in Veterans With SUD/PTSD in a Residential Treatment Program
Brief Title: OSA PAP Treatment for Veterans With SUD and PTSD on Residential Treatment Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3623-R; 1I01RX003623-01 (NIH)
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Post Traumatic Stress Disorder; Obstructive Sleep Apnea; Substance Use Disorder; Residential Treatment Program
Keywords: Veteran; PTSD; Obstructive Sleep Apnea; Substance Use Disorder; PAP Treatment; Residential Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Apnea, Obstructive; Substance-Related Disorders | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: The investigators aim to examine the effects of PAP treatment on Veterans with PTSD and SUD on a 28-day residential unit. The investigators are proposing a randomized controlled study comparing two groups: an early intervention PAP treatment group receiving PAP treatment while on the residential unit, compared to a waitlist control group who will receive PAP treatment at 3-months post-discharge follow-up.
Who Masked: Outcomes Assessor
Masking Description: All assessors will be blinded to treatment condition to minimize bias in outcome assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAP Treatment on SARRTP Unit (Experimental): Veterans will receive Positive Airway Pressure device while on the 28-day SARRTP Unit.
  Interventions: Device: Positive Airway Pressure Device
- Waitlist Control (No Intervention): Veterans will not receive PAP device until after 3-month Follow Up.

INTERVENTIONS:
Device: Positive Airway Pressure Device — Each PAP treatment initiation meeting will include 1) mask fitting; 2) psycho-education to what to expect and reviewing PAP machine problem solving; and 3) setting up correct PAP treatment (e.g., auto PAP or in rare conditions, bi-level PAP).
  Other Names: PAP; CPAP; Auto-PAP
  Arms: PAP Treatment on SARRTP Unit

SUMMARY:
Substance use disorder (SUD) and posttraumatic stress disorder (PTSD) frequently co-occur and having both disorders is associated with greater psychological and functional impairment than having either disorder alone. This is especially true in residential settings where both disorders are more severe than outpatient settings. Obstructive sleep apnea (OSA) is highly comorbid with both disorders and untreated OSA is associated with worse functional impairment across multiple domains, worse quality of life, worse PTSD, higher suicidal ideation, and higher substance use and relapse rates. Treating OSA with evidence-based positive airway pressure (PAP) in Veterans with SUD/PTSD on a residential unit is a logical way to maximize treatment adherence and treatment outcomes. This study compares OSA treatment while on a SUD/PTSD residential unit to a waitlist control group. The investigators hypothesize that treating OSA on the residential unit, compared to the waitlist control, will have better functional, SUD, and PTSD outcomes.

DETAILED DESCRIPTION:
Substance use disorder (SUD) and posttraumatic stress disorder (PTSD) frequently co-occur and having one condition worsens the course of the other. Individuals with both disorders exhibit worse functioning across a number of domains than individuals with either disorder alone. This is especially true in residential settings where both disorders are more severe than outpatient settings. Compared to Veterans with a single disorder, Veterans with SUD/PTSD also are more likely to have suicidal ideation and to have attempted suicide. Examining treatable conditions that are associated with improved SUD and PTSD outcomes, such as obstructive sleep apnea (OSA), can maximize treatment efficacy for Veterans at a critical time in recovery.

OSA is highly comorbid with both PTSD and SUD with upwards of 67 to 83% of Veterans with SUD or PTSD also having OSA. Further, untreated OSA is associated with worse functional impairment across multiple domains, worse quality of life, worse PTSD, and higher substance use and relapse rates. Importantly, untreated OSA also contributes to higher suicide attempts and completion. Positive airway pressure (PAP) is the gold standard treatment for OSA with large effects on multiple domains of functioning, quality of life, PTSD symptoms, physical functioning, lower depression, and better emotional coping. Unfortunately, screening and treating Veterans for OSA is not a part of clinical practice for SUD or PTSD treatment; as such the average wait time for individuals to get PAP therapy is upward of two years. Despite the widespread dissemination of knowledge regarding the detrimental effects of untreated OSA and the incredible effectiveness of PAP treatment, OSA is rarely screened for or treated in patients with SUD or PTSD, with approximately 80% to 90% of Veterans with OSA remaining undiagnosed and untreated.

Methodology.

The investigators aim to examine the effects of PAP treatment on Veterans with PTSD and SUD on a 28-day residential unit. The investigators are proposing a randomized controlled study comparing two groups: an early intervention PAP treatment group receiving PAP treatment while on the residential unit, compared to a waitlist control group who will receive PAP treatment at 3-months post-discharge follow-up. Participants will be 194 male and female Veterans on the residential SUD and PTSD unit with SUD, PTSD, and OSA. The primary aim is to determine the relative efficacy of PAP treatment on the SUD/PTSD unit, as compared to waitlist control, in reducing problematic substance use, PTSD symptoms, and suicidal ideation, while improving functioning among Veterans with comorbid SUD/PTSD at 3-months post-treatment follow-up. The investigators will also compare PAP adherence rates on PTSD/SUD/functioning outcomes within the PAP treatment group (3-months). Finally, the investigators plan on comparing adherence rates between the two treatment groups at the 6-months post-treatment follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* a Veteran of the U.S. military or Reserve/National Guard member
* at least 18 years of age
* have an AHI 5 per hour
* experienced trauma that occurred in childhood or adulthood; at least one month post-trauma
* have current DSM-5 diagnoses of SUD via SCID-SUD module with a minimum 20 days of substance use in the last 90 days (Timeline Follow-back)
* Full PTSD diagnosis via clinician administered PTSD scale
* are literate in English
* are on the PTSD track of the SARRTP unit
* are capable of giving informed consent

Exclusion Criteria:

* have central sleep apnea (AHI >=5 and > 50% central apneas)
* arrives on the SARRTP unit already using a PAP device (Veteran's previously diagnosed with OSA, but not using PAP therapy will be eligible)
* the SARRTP medical staff advises against the study based on medical history and physical examination; d) history of severe cognitive impairment (via MOCA < 26)
* history of psychosis or mania independent of substance use will be excluded because the presence of these disorders can impede therapy progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, Post-SARRTP Unit (28 Days), 3-Month Follow up (90 Days)
  Change in functional impairment across multiple domains. The WHODAS 2.0 is a 36-item questionnaire that assess functional impairment across 5 subscales: cognitions (understanding and communicating), mobility, self-care getting along with others, household responsibilities, work responsibilities, and community participation.
Change in Timeline Follow-Back (TLFB) % days drinking/using in last 90 days | Baseline, 3-Month Follow up (90 Days)
  Examining change in percentage of substance use in the past 90 days.
Change in Clinician Administered PTSD Scale (CAPS-5) | Baseline, Post-SARRTP Unit (28 Days), 3-Month Follow up (90 Days)
  Change in PTSD symptom severity will be assessed using CAPS-5 in the past month. The CAPS-5 is a 30-item structured interview.
Change in The Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, Post-SARRTP Unit (28 Days), 3-Month Follow up (90 Days)
  Change in suicidal ideation severity using the C-SSRS. The C-SSRS is a standardized 8-point clinician-administered suicidal rating system designed to track suicidal adverse events across a treatment trial and covering the wide spectrum of suicidality

SECONDARY OUTCOMES:
PAP adherence rates | 3-Month Follow up (90 Days)
  Examining average number of nights used positive airway pressure is use over the last 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Colvonen, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No